CLINICAL TRIAL: NCT04128033
Title: Impact of the Puncture of the RP6 Point on the Ampliation and Injuries of the Perineum During Childbirth
Acronym: PELVPUNCTURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-A03070-55
Record Dates: First submitted 2019-10-14; First posted 2019-10-16 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Perineum; Injury
Keywords: acupuncture; perineum injury; delivery
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Monocentric, randomized, simple blinded, controlled study
Who Masked: Participant
Masking Description: Participant doesn't know if the point punctured is the experimental or the placebo point.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- puncture of the RP6 point (Experimental): The acupuncturist midwife, who does not perform the delivery herself, punctures the RP6 point at the time of the expulsive efforts.
  Interventions: Other: Puncture of the RP6 point
- puncture of the placebo point (Placebo Comparator): The acupuncturist midwife, who does not perform the delivery herself, punctures the placebo point at the time of the expulsive efforts.
  Interventions: Other: Puncture of the placebo point

INTERVENTIONS:
Other: Puncture of the RP6 point — Puncture of RP6 "San Yin Jiao" point, located just behind the posterior edge of the tibia 3 cm above the end of the inner malleolus.
  Arms: puncture of the RP6 point
Other: Puncture of the placebo point — Puncture of a placebo point "outside the meridian", with no effect
  Arms: puncture of the placebo point

SUMMARY:
During the study period, any patient who enters labour and reports to the maternity ward and meets the inclusion and non-inclusion criteria is offered to participate in the study by the midwife acupuncturist present.

After signing the informed consent, a numbered envelope with the randomization arm is assigned to the patient. The acupuncturist midwife does not perform the delivery herself. At the time of the expulsive efforts, she punctures the point drawn at random. The patient's participation in the study ends when she leaves the labour room after the birth.

DETAILED DESCRIPTION:
During the study period, any patient who enters labour and reports to the maternity ward and meets the inclusion and non-inclusion criteria is offered to participate in the study by the midwife acupuncturist present. She's responsible for explaining the purpose and practicalities of the study orally and issues a written information document. The information provided is the same regardless of the midwife present. If she agrees to participate in the study, the patient signs the consent form.

After signing the informed consent, a numbered envelope with the randomization arm is assigned to the patient. The acupuncturist midwife does not perform the delivery herself. At the time of the expulsive efforts, she punctures the point drawn at random. She collects the clinical Research Form from the time the patient signs the consent form until she leaves the labour room after the birth.

The patient's participation in the study ends when she leaves the labour room after the birth. No further follow-up is planned.

ELIGIBILITY:
Inclusion Criteria:

* primiparous or multiparous women who have never given birth vaginally
* term patients (after 37 weeks of amenorrhea)
* patients delivering a fetus in cephalic presentation
* patients speaking and understanding French.

Exclusion Criteria:

* patients suspected of having a fetal macrosomy (greater than the 97th percentile) on the last ultrasound
* patients with twin pregnancies
* excised patients
* patient who has made an acupuncture preparation during pregnancy
* patients with fetal death in utero
* patients requiring medical termination of pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Rate of intact perineum after childbirth | immediately after childbirth
  Rate of intact perineum after childbirth

SECONDARY OUTCOMES:
Rate of simple perineal tears | immediately after childbirth
  lesion of the skin, vaginal mucosa, connective tissue, or sometimes the superficial muscle plane
Rate of complete perineal tears | immediately after childbirth
  Sphincter damage to the anus
Rate of complicated complete perineal tears | immediately after childbirth
  Damage to the anal mucosa
Rate of episiotomies performed | immediately after childbirth
  Rate of episiotomies performed

CONTACTS AND LOCATIONS:
Overall Officials: Berangère BC CANON, MD, Study Director — Centre Hospitalier Sud Francilien
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France